CLINICAL TRIAL: NCT04262830
Title: CATCH-HF: Cardiotoxicity Assessment Through Comprehensive Heart Imaging to Predict Heart Failure
Brief Title: Cardiotoxicity Assessment Through Comprehensive Heart Imaging to Predict Heart Failure
Acronym: CATCH-HF
Status: Recruiting | Type: Observational
Sponsor: Hari Narayan (Other)
Responsible Party: Sponsor-Investigator, Hari Narayan, Assoc Physician Dipl, University of California, San Diego
Organization: University of California, San Diego (Other)
Other Study IDs: 181758
Record Dates: First submitted 2019-11-04; First posted 2020-02-10 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Cardiotoxicity; Pediatric Cancer; Heart Failure
MeSH Terms: conditions — Cardiotoxicity; Neoplasms; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All Study Participants: This is an observational study where all study participants are within a single group.
  Participants will have testing performed at baseline and again at follow-up >= 3 years after the initial assessment.
  Interventions: Diagnostic Test: Cardiac magnetic resonance imaging (MRI); Other: Accelerometer physical activity monitoring

INTERVENTIONS:
Diagnostic Test: Cardiac magnetic resonance imaging (MRI) — Cardiac magnetic resonance imaging will be performed to evaluate cardiac remodeling, function, and tissue characteristics
Other: Accelerometer physical activity monitoring — Measurement of physical activity using hip-worn accelerometer.

SUMMARY:
Anthracycline chemotherapies (e.g. doxorubicin, daunorubicin) are commonly given to treat pediatric cancer, and carry a risk of cardiotoxicity. Over the long term, children who receive these therapies have an increased risk of heart failure and early cardiovascular death. However, current strategies for identifying patients who are at risk prior to the development of significant changes in heart function are limited. This study will focus on imaging markers of cardiac injury and dysfunction with the goal of developing improved diagnostic tests and treatment strategies.

DETAILED DESCRIPTION:
Anthracycline chemotherapies (e.g. doxorubicin, daunorubicin) are commonly given to treat pediatric cancer, and carry a risk of cardiotoxicity. Over the long term, children who receive these therapies have an increased risk of heart failure and early cardiovascular death. However, current strategies for identifying patients who are at risk prior to the development of significant changes in heart function are limited. This study will focus on imaging markers of cardiac injury and dysfunction with the goal of developing improved diagnostic tests and treatment strategies.

Cardiac remodeling, function, and tissue characteristics will be examined using cardiac MRI in combination with other research assessments to assess the cardiotoxic effects of cancer therapy. Analyses will be performed in a cohort of adolescents and young adults with a history of childhood cancer.

ELIGIBILITY:
Inclusion Criteria:

* English and Spanish speaking male and female subjects, ages 13-39 years old
* Diagnosis of cancer at age <22 years
* Previously treated with anthracyline therapy for cancer, with diagnosis at least two years prior.

Exclusion Criteria:

* Patients who have a contraindication to cardiac MRI, including the presence of non-MRI compatible metallic implants.
* Medical, psychiatric, and/or social disorder that would prevent successful completion of planned study testing or would preclude the subject from undergoing the cardiac MRI without anesthesia.
* Patients with a history of congenital heart disease (more significant than a history of patent foramen ovale or patent ductus arteriosus).
* Pregnancy (at the time of enrollment).

Ages: 13 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Long-term childhood cancer survivors treated with anthracyline therapy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (LVEF) | 3 - 5 years
  LVEF is an assessment of left ventricular global systolic function.

CONTACTS AND LOCATIONS:
Overall Officials: Hari Narayan, MD, Principal Investigator — University of California San Diego, Rady Children's Hospital
Locations (1):
- Rady Children's Hospital, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided